CLINICAL TRIAL: NCT03855683
Title: Transdiagnostic Interventions for Emotional Disorders
Brief Title: Stress, Anxiety, and Mood Group Therapy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Social distancing regulations related to COVID19.
Sponsor: Palo Alto University (Other)
Responsible Party: Principal Investigator, Stacie Warren, Ph.D., Principal Investigator, Palo Alto University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-061
Record Dates: First submitted 2019-02-10; First posted 2019-02-27 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Depressive Disorders; Anxiety Disorders
Keywords: depression; anxiety
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group therapy (Unified Protocol) (Experimental): Participants experiencing stress, anxious, and/or depressive symptoms will receive 8 sessions of Unified Protocol for Emotional Disorders lasting for 90 minutes each. Includes psycho-education about (mal)adaptive emotion regulation, cognitive and behavioral tools to reduce symptoms of stress, anxiety, and/or depression.
  Interventions: Behavioral: Unified Protocol for The Treatment of Emotional Disorders

INTERVENTIONS:
Behavioral: Unified Protocol for The Treatment of Emotional Disorders — Unified Protocol (UP) is is an 8-week intervention designed to specifically benefit individuals who report co-occurring symptoms of anxiety, stress, and mood by providing them with psychoeducation regarding (mal)adaptive emotion regulation, as well as with skills for effectively responding to stress. UP is based on a cognitive-behavioral framework and uses cognitive and behavioral therapy techniques. Each session of UP group therapy is 90 minutes in duration. Sessions themselves generally include a review of homework and previously discussed concepts, introduction of new material, and in-session discussions/activities.

SUMMARY:
The purpose of this study is to identify cognitive mechanisms that might facilitate treatment response for individuals experiencing depression and/or anxiety. The Stress, Anxiety, and Mood group helps individuals experiencing symptoms of stress, anxiety, and mood by providing concrete coping skills to regulate emotions, to let go of negative thoughts, and build courage to talk to others about tough topics. Groups meet for 8 weeks, with sessions lasting 90 minutes each. In addition to group therapy, you will be asked to complete some computerized and paper and pencil-based tasks.

If you are interested in learning more, please contact us at 650-417-2000 ext. 3642 or paloalto.study@gmail.com. All inquiries will be kept strictly confidential.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify specific patterns of executive function impairment that distinguish affective and cognitive symptoms in anxious and/or depressed patients.

II. Identify specific components of executive function that predict Unified Protocol treatment response. This will set up subsequent cognitive intervention studies targeting those components.

The phone screen includes a confidentiality statement explaining how their information will be kept confidential, demographic questions, and questions regarding the participants' medical and psychiatric history, and current psychological state. Responses to these questions will be used to determine if the individual meets inclusion criteria to engage in the study. If the participant meets study eligibility criteria, he/she will be invited to an informational session not exceeding two and a half hours at Dr. Warren's lab, which involves an explanation the project, informed consent, some questionnaires, and a diagnostic clinical interview. Also during the first visit, participants will be informed of the upcoming visits and the types of activities they will be asked to engage in for the purposes of this study. During a second visit, subjects will undergo cognitive testing designed to measure set shifting, working memory updating, cognitive inhibition, processing speed, general intelligence, and attentional control. These tests will be administered at Dr. Warren's lab and will not exceed two and a half hours. The remainder of the study visits will involve an 8-week, cognitive-behavioral group therapy titled "Unified Protocol," to take place at the Gronowski Clinic. Treatment groups will be facilitated by Dr. Warren and co-facilitated by trained graduate students selected by Dr. Warren.

ELIGIBILITY:
Inclusion Criteria:

* Normal color vision
* Ability to travel to Palo Alto University
* Experiencing symptoms of stress, anxiety, and/or depression

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Level of depression as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Mood and Anxiety Symptom Questionnaire- Anhedonic Depression subscale
Level of intolerance of uncertainty as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Intolerance of Uncertainty Questionnaire
Level of rumination and reflection as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Rumination Reflection Questionnaire
Level of anxious arousal as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Mood and Anxiety Symptom Questionnaire- Anxious Apprehension subscale
Level of anxious apprehension as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Penn State Worry Questionnaire
Level of alcohol use as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Alcohol Use Disorders Identification Test
Level of positive and negative emotions as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  The Positive and Negative Affect Schedule
Level of behavioral regulation and metacognition as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Behavioral Regulation Index and Metacognition Index
Level of trait mood as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Trait Meta-Mood Scale.
Level of emotion regulation as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Emotion Regulation Questionnaire
Level of mental imagery as measured by the following questionnaire: | The change from baseline and post-treatment, approximately 8 weeks after baseline
  Questionnaire of Mental Imagery
Level of cognitive functioning via neuropsychological testing session | Baseline
  Objective assessment of cognitive strengths and weaknesses

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Warren, PhD, Principal Investigator — Palo Alto University
Locations (1):
- Palo Alto University, Los Altos, California, United States

IPD SHARING:
Plan to Share IPD: No